CLINICAL TRIAL: NCT04904029
Title: Validation and Implementation of a Digital Assessment Routing Tool (DART) as an Alternative to Physiotherapy-led Remote Triage for Musculoskeletal Disorders: Protocol for a Pilot Randomised Crossover Non-inferiority Trial
Brief Title: Digital Assessment Routing Tool (DART): Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Optima Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: OH_QMUL_DART-Pilotstudy
Record Dates: First submitted 2021-03-19; First posted 2021-05-27 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Diseases or Conditions
Keywords: Musculoskeletal disorders; Physiotherapy; Web-based tool; Telehealth; Musculoskeletal; DART; Digital tool; Triage; Remote triage; Musculoskeletal management; Musculoskeletal triage; Clinical algorithm; Digital assessment routing tool; MSK; MSD; Telephone triage
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Pilot study to inform a pilot randomised, double-blinded, crossover, non-inferiority trial with two arms (to account for order effects).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator will be blinded for group intervention and outcomes data-analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Digital Assessment Routing Tool (DART) 2. Physiotherapy-led remote triage (Experimental): Participants complete the Digital Assessment Routing Tool (DART), which is followed by physiotherapy-led remote triage with the usual care clinician.
  Interventions: Other: Digital Assessment Routing Tool [DART]; Other: Physiotherapy-led remote triage (usual care)
- 1. Physiotherapy-led remote triage 2. Digital Assessment Routing Tool (DART) (Experimental): Participants complete their physiotherapy-led remote triage with the usual care clinician, which is followed by the Digital Assessment Routing Tool.
  Interventions: Other: Digital Assessment Routing Tool [DART]; Other: Physiotherapy-led remote triage (usual care)

INTERVENTIONS:
Other: Digital Assessment Routing Tool [DART] — DART is a first contact web-based and mobile health system that uses clinical algorithms to triage patients and recommend management pathways. Participants complete an online web-based questionnaire that follows a clinical reasoning process commonly observed in face-to-face physiotherapy consultations. Based on the participant's answers, the clinical algorithm generates sets of questions, leading up to a triage disposition with recommended management pathway. The triage outcomes with management pathways are classified;
  1. Medical care
     * A&E referral
     * Urgent GP
     * Routine GP
     * Consultant review
  2. Physiotherapy care
     * Post-fracture or surgery physiotherapy
     * Physiotherapy referral
     * Physiotherapy referral plus psychosocial support
  3. Self-management
     * Self-management with SOS
     * Continue self-management advice
Other: Physiotherapy-led remote triage (usual care) — Participants will receive usual physiotherapy-led remote triage services by a registered health care professional. This service is either a telephone or video consult and includes any diagnostic procedure (e.g. patient history, remote assessments) and treatment, such as management advise or home-based exercise therapy. Participants may seek help elsewhere or opt-out the study at any point, which will not affect their usual physiotherapy-led remote care

SUMMARY:
In the pilot study, we aim to explore trial design, assess procedures, and collect exploratory data to inform the design of a future Randomised Controlled Trial.

The intervention involves a Digital Assessment Routing Tool (DART) that provides triage outcomes with recommended management pathways for participants with musculoskeletal problems. Participants complete DART either before or after their consultation with usual care clinicians (Physiotherapy-led remote triage). The triage outcome dispositions between DART and usual care clinicians will be compared.

A panel will be formed to provide consensus on disagreements that may result in adverse triage outcomes, as well as on a sample of agreements between DART and usual care clinicians.

DETAILED DESCRIPTION:
The Digital Assessment Routing Tool (DART) is a first-contact web-based and mobile health system that uses clinical algorithms to triage patients with musculoskeletal disorders and recommend management pathways. This is achieved by completing an online web-based questionnaire that follows a clinical reasoning process commonly observed in face-to-face physiotherapy consultations. Based on the participant's answers, the clinical algorithm will generate sets of questions, leading up to a final triage disposition with a recommended management pathway. The triage outcomes with recommended management pathways are classified as follows;

1. Medical care

   * A&E referral
   * Urgent GP
   * Routine GP
   * Consultant review
2. Physiotherapy care

   * Post-fracture or surgery physiotherapy
   * Physiotherapy referral
   * Physiotherapy referral plus psychosocial support
3. Self-management

   * Self-management with SOS
   * Continue self-management advice

The usual care clinician, providing physiotherapy-led remote triage, will follow their clinical reasoning and proceed with the consultation as usual. The participants will receive both the DART assessment and usual care remote triage (crossover design). Patient care will not change (except time taken to reach a decision) as its a crossover design and only the clinician assessment will count. Note, participants will be randomised in two arms (DART, PT-remote triage or reversed) to account for order effects.

Outcomes will be collected at a single time point (Visit 1).

Post data collection, a panel consisting of researchers, physiotherapists and clinical leaders with a minimum of 5 years' experience in musculoskeletal health will provide consensus on all the disagreements between DART and physiotherapy-led remote triage that can result in adverse triage outcomes;

* Physiotherapy care or self-management when it should have been urgent medical care (A&E referral or urgent GP).
* Self-management when it should have been either physiotherapy care or medical care and harm could result.
* Routine care when it should have been urgent care and harm could result.

In addition, random samples of triage outcomes will be assessed to decide whether they were the most appropriate outcome.

ELIGIBILITY:
Inclusion Criteria:

* A current musculoskeletal injury for which they are seeking treatment
* Over 18 years old
* Able to read and speak English
* Live in the UK
* Able to access the internet

Exclusion Criteria:

* Cognitive impairments or learning disabilities that limits the participants to follow study- related procedures
* Unwillingness or inability to follow protocol-related procedures
* Optima Health employees
* Has an assessment from a health care professional for the same condition within the last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
The agreement rate between triage outcomes with management pathways from physiotherapy-led and DART triage assessments. | Immediately after the intervention.
  The primary outcome measure will be the agreement rate of triage decisions made by both the clinician and the Digital Assessment Routing Tool (DART). The possible triage outcomes with management pathways are classified in three categories, namely 1) Medical care, 2) Physiotherapy care, and 3) Self-management.
  1. Medical care
     * A&E referral
     * Urgent GP
     * Routine GP
     * Consultant review
     * Physiotherapy care
  2. Post-fracture or surgery physiotherapy
     * Physiotherapy referral
     * Physiotherapy referral plus psychosocial support
     * Self-management
  3. Self-management
     * Self-management with SOS
     * Continue self-management advice

OTHER OUTCOMES:
Proportion of participants identified, shown interest to participate, and recruited to the study. | Through study completion, an average of 3 months.
  Participants drop-out rates at each stage of the trial (and where possible reasons for dropping out) will be collected. A pre-defined criterion of 50% and 95% will be considered satisfactory for the proportion of identified participants recruited and retained, respectively.
The number of errors reported in randomisation, allocation concealment, blinding or data collection. | Immediately after the intervention.
  System process outcomes include errors reported in randomisation, allocation concealment, blinding or data collection. Any evidence for selection bias or other sources of bias will be explored.
Time burden (in minutes) of interventions. | Immediately after the intervention.
  The overall time burden (in minutes) will be estimated from initial participant contact to first treatment, along with any treatment delay due to the additional time required to perform research procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Morissey, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Haydock Medical Centre, St Helens, Herts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lowe C, Sephton R, Marsh W, Morrissey D. Evaluation of a Musculoskeletal Digital Assessment Routing Tool (DART): Crossover Noninferiority Randomized Pilot Trial. JMIR Form Res. 2024 Jul 30;8:e56715. doi: 10.2196/56715. PMID 39078682
- [Derived] Lowe C, Hanuman Sing H, Marsh W, Morrissey D. Validation of a Musculoskeletal Digital Assessment Routing Tool: Protocol for a Pilot Randomized Crossover Noninferiority Trial. JMIR Res Protoc. 2021 Dec 13;10(12):e31541. doi: 10.2196/31541. PMID 34898461

DOCUMENTS (1):
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT04904029/ICF_000.pdf